CLINICAL TRIAL: NCT04616287
Title: Self in Dementia With Lewy Bodies: a Behavioral and Multimodal Neuroimaging Study
Brief Title: Self and Autobiographical Memory in Dementia With Lewy Bodies and Alzheimer Disease: a Behavioral and Multimodal Neuroimaging Study
Acronym: SELF-MCL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 7942
Record Dates: First submitted 2020-11-02; First posted 2020-11-04 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Dementia With Lewy Bodies; Alzheimer Disease; Self; Autobiographical Memory; Insular Cortex
MeSH Terms: conditions — Lewy Body Disease; Alzheimer Disease | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- dementia with Lewy bodies (Experimental)
  Interventions: Other: Neuropsychological assessment and Multimodal brain MRI
- Alzheimer disease (Active Comparator)
  Interventions: Other: Neuropsychological assessment and Multimodal brain MRI
- healthy elderly subjects (Sham Comparator)
  Interventions: Other: Neuropsychological assessment and Multimodal brain MRI

INTERVENTIONS:
Other: Neuropsychological assessment and Multimodal brain MRI — Neuropsychological assessment and Multimodal brain MRI

SUMMARY:
The present project aims at exploring different components of Self-consciousness or 'the Self', such as autobiographical memory, self-concept and subjective sense of Self, in dementia with Lewy Bodies (DLB) compared to Alzheimer's disease and to normal ageing. Anatomical substrates will be studied in multimodal imaging, in terms of volume, anatomical and functional connectivity. We expect to find an alteration of the different components of the Self, consecutive to insular dysfunction, a key region within cerebral networks of self-consciousness, which is damaged early in the course of the disease.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for all participants:

* Male or female aged between 60 to 80, at the inclusion visit
* Right-handed
* Must be affiliated to a social health insurance protection scheme
* Must be able both to understand the objectives and risks related to the study and to give a dated and signed informed consent
* Fluency in French
* At least 9 years of formal education

Inclusion criteria for group of dementia with Lewy bodies:

* Subject meeting McKeith et al. criteria (2017)
* Subject with prodromal dementia with Lewy bodies meeting the DSM-V Mild Cognitive Impairment criteria (2013)
* Subject with prodromal or mild dementia with Lewy bodies with an ≤ 20 MMSE score
* Availability of a caregiver for the inclusion visit

Inclusion criteria for group of Alzheimer disease:

* Subject meeting Dubois et al. criteria (2014)
* Subject with prodromal or mild Alzheimer disease with an ≤ 20 MMSE score
* Availability of a caregiver for the inclusion visit

Inclusion criteria for healthy elderly:

* Subject must be matched with patients in terms of age, gender and educational level
* Absence of any cognitive complaint
* Autonomy must be preserved

Exclusion Criteria:

Subjects with significant neuropsychiatric comorbidities

* Abnormal neurological examination
* Sensory impairment that may significantly interfere with testing
* Contraindication to MRI
* Claustrophobia
* Heavy psychotropic drug treatment
* Excessive and regular consumption of alcohol
* Subject in period of exclusion (determined by a previous or ongoing study)
* Inability to give the subject informed information
* Subject under judicial protection
* Subject under tutorship or guardianship

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-10-23 (Actual)

PRIMARY OUTCOMES:
Neuropsychological assessment | months 3
Multimodal brain MRI | months 3

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie PHILIPPI, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tisserand A, Philippi N, Botzung A, Blanc F. Me, Myself and My Insula: An Oasis in the Forefront of Self-Consciousness. Biology (Basel). 2023 Apr 14;12(4):599. doi: 10.3390/biology12040599. PMID 37106799